CLINICAL TRIAL: NCT06696469
Title: Feasibility and Reliability of Using BeCureTM Virtual Reality in the Evaluation of Upper Extremity Motor Functions in Patients With Stroke
Brief Title: Feasibility and Reliability of Using BeCureTM Virtual Reality in Patients With Stroke
Acronym: cros-sectional
Status: Recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Şehim Kutlay, Professor Doctor, Ankara University
Other Study IDs: I06-427-24
Record Dates: First submitted 2024-11-14; First posted 2024-11-20 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Stroke Patients
Keywords: upper limb motor functions; stroke; virtual reality
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient group: Post-stroke patients
  Interventions: Diagnostic Test: Feasibility and reliability of using BeCureTM Virtual Reality in the evaluation of upper extremity motor functions in stroke patients

INTERVENTIONS:
Diagnostic Test: Feasibility and reliability of using BeCureTM Virtual Reality in the evaluation of upper extremity motor functions in stroke patients — The applicability and reliability of virtual reality systems are important factors to consider. Based on this, this study aimed to investigate the feasibility of using BeCureTM virtual reality in the evaluation of upper extremity functions after stroke.The feasibility of using BeCureTM virtual reality in stroke patients will be determined according to the System Usability Scale (SUS) score.The safety of the use of BeCureTM virtual reality in stroke patients will be assessed with a patient feedback questionnaire. The relationship between the use of BeCureTM virtual reality and cognitive functions in stroke patients will be determined by the Montreal Cognitive Assessment Scale and Mini Mental State Examination.It was aimed to examine the effects of demographic characteristics, accompanying cognitive disorders and upper extremity motor disorders that may affect the evaluation and response to treatment on virtual reality applications.

SUMMARY:
The aim of this study is to demonstrate the feasibility and reliability of using virtual reality-based BeCureTM in the assessment of upper extremity motor functions in stroke patients.It is necessary to define the appropriate patient profile for the evaluation of upper extremity motor functions in stroke patients with virtual reality method. We aimed to examine the effects of demographic characteristics, accompanying cognitive disorders and upper extremity motor disorders that may affect the evaluation and response to treatment on virtual reality applications. Therefore, BeCure TM virtual reality system can be feasibly used in the evaluation and rehabilitation of stroke patients.

DETAILED DESCRIPTION:
Various motor disorders such as muscle weakness, decreased range of motion and coordination frequently occur after stroke. With the deterioration of fine and gross motor skills, especially in the upper extremities, the individual has difficulty in performing daily life activities and becomes dependent. With the introduction of advanced technologies in the field of rehabilitation, robotic rehabilitation and virtual reality applications have become widespread in our country as well as all over the world in recent years. Virtual reality allows for objective and quantitative assessment on the one hand and contributes to the rehabilitation process through serious games on the other. Virtual reality applications are frequently used in the evaluation of upper extremity functions after neurological diseases (e.g. stroke, cerebral palsy, multiple sclerosis). Virtual reality systems can allow skill-oriented exercises to be performed in a fun and safe environment while keeping the patient's interest and motivation at a high level. Thus, they can also provide access to the intensity and quality of exercise required to increase neuroplasticity. In the literature, there are studies showing that virtual reality technologies improve motor function in stroke patients. Patients with stroke may develop cognitive disorders such as attention deficit, apraxia, visual-spatial perception, neglect and memory, motor and sensory disorders, balance and posture disorders, speech and language disorders such as aphasia-dysarthria. It is necessary to define the appropriate patient profile in the evaluation of upper extremity motor functions in stroke patients with virtual reality method. The aim of this study was to examine the effects of demographic characteristics, accompanying cognitive disorders, and upper extremity motor disorders on virtual reality applications that may affect the evaluation and response to treatment. Therefore, BeCure TM virtual reality system can be feasibly used in the evaluation and rehabilitation of stroke patients.The study will be conducted in the Physical Medicine and Rehabilitation Clinic of Ankara University Faculty of Medicine Cebeci Hospital between 22.06.2024 and 22.06.2026. Volunteers who develop hemiplegia after stroke and healthy volunteers will be included in the study. Volunteers will be evaluated by Dr. Funda YAŞAR using the patient follow-up form (attached).Accordingly, sociodemographic information, history of previous computer or touchscreen phone use and gaming experience, time of diagnosis and type of lesion (ischemic or hemorrhagic), affected body half, background and dominant hand status of all volunteers, and accompanying cognitive impairments will be determined. In the subsequent physical examination, the state of consciousness, orientation and cooperation will be evaluated and mini mental test will be applied.The Mini Mental Test (MMT) is a screening test used to rapidly determine general cognitive status. The test consists of orientation, recording, attention and calculation, recall and language sections and is scored out of 30 points.The Montreal Cognitive Assessment (MoCA) scale was planned to be used to assess cognitive functions.The MoCA was developed as a rapid screening test for mild cognitive impairment. The test is a 30-point test assessing visual/spatial-administrative functions, naming, memory, attention, language, abstract thinking, recall and orientation.A score of 21 and above is considered normal.This study will include participants who can understand commands.Brunnstrom motor staging will be used for motor evaluation of the patients. This staging system consists of 3 sections: upper extremity, hand and lower extremity. The sections are graded from 1-7. A higher grade indicates a better motor stage. Volunteers with Brunnstrom upper extremity stage 3 and above will be included in the study. The Fugl-Meyer Rating Scale (FMRS) was planned to be used to assess upper extremity (UE) motor function.In our study, the UE motor function section of the FMDI will be used. UE motor function is evaluated in 4 subheadings. The total score is 66 points (0-66 points) including UE 36, wrist 10, hand 14 and coordination speed 6 points. Higher scores indicate better motor function. In UE, the motor function section is assessed in approximately 30 minutes.The Modified Ashworth Scale will be used to assess spasticity in stroke survivors.Accordingly, participants with spasticity grade 3 and above in the upper extremity will be excluded from the study because it will prevent movement in the upper extremity.The Barthel activities of daily living index is an assessment scale used to measure an individual's performance in activities of daily living.The aim of this scale is to determine to what extent the patient can perform these actions independently without any physical or verbal assistance.The 9-hole peg test assesses manual dexterity, strength, visual attention, depth perception, sensory perception and motor coordination.BIT (Behavioral Inattention Test) was planned to be used to determine the Neglect Syndrome. The patient will be given a test consisting of dividing the line in half, copying the figure and shape, drawing the depicted shape, canceling the star, drawing over the line, canceling the letter. The classical score will be 146 and the behavioral score will be evaluated out of a total of 81 points.The System Usability Scale (SUS) is a simple, ten-item Likert scale of subjective evaluations of usability.In short, it is a standardized questionnaire to measure users' satisfaction with a product or system. Developed in 1986 by John Brooke for usability evaluation. In short, it is a standardized questionnaire to measure users' satisfaction with a product or system. At the same time, a score between 0-100 can be obtained with SUS. When calculating the exact score, 1 is subtracted from the given value of items 1, 3, 5, 7 and 9 (odd numbered and positive opinion). The scores for items 2, 4, 6, 8 and 10 (items with negative opinions) are subtracted from 5. The SUS score can then be found by adding them all together and multiplying this sum by 2.5 to complete the 0-100 range.After the section including questioning and physical examination is completed, the virtual reality application phase will be started for volunteers who meet the specified inclusion criteria. The volunteers included in the study will be positioned in a sitting position at the edge of the table. BecureTM virtual reality-based Leap Ball game will be played on a laptop computer. Leap Ball is a game that can be applied in neurological diseases such as cerebral palsy, multiple sclerosis, stroke, etc. and all hand diseases. It is aimed to perform flexion/extension, adduction/abduction movements of the wrist and fingers with Leap Ball. In this application, the volunteer will be practiced 2 times and then the game will be started. In this application, the upper extremity and hand movements of the person will be reflected on the computer screen through the motion sensor (Leap Motion Controller), which is positioned on the table on the laptop screen and does not touch the volunteer. The game will start when the start button is pressed. When the patient hears the command 'hold the ball' with the instruction sound, he/she will grasp the ball and take the ball to the open hole. With the 'drop the ball' command, the patient will drop the ball into the hole. If the target number of balls enters the hole within the specified time, the game will end successfully. After the game, the completion time will be displayed on the screen. Leap ball virtual reality application takes approximately 15 minutes. In healthy volunteers who are similar in terms of age and gender, the game will be applied in both dominant and non-dominant hand, and in the group of volunteers who had a stroke, the game will be played with the hemiplegic side. The game will be repeated in the same way 7 days after the first evaluation. Patients treated in the virtual reality treatment unit will be evaluated 2 times in total. The first evaluation will be done in the process of getting used to the system. The 2nd evaluation will be done 1 week later. Subsequently, the patient will be asked to fill out the SUS scale and patient feedback questionnaire, which evaluates the applicability and reliability. The patient feedback questionnaire will be filled out by Dr. Funda Yaşar, who played the game, after the 2nd evaluation, by face-to-face interviews with the patients to evaluate their thoughts about the game system. MMT, MoCA, Nine hole peg test was planned to be performed in healthy volunteers. Dominant and non-dominant extremities will be evaluated with the Nine Hole peg test. A virtual reality game will be played on the dominant and non-dominant extremity and the time to finish the game will be recorded. SUS and patient feedback questionnaire will be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with stroke according to the World Health Organization with an age range of 18-80 years
2. Patients with subacute to chronic stroke
3. Patients who can understand commands
4. Patients with sitting balance
5. Patients with a first stroke attack
6. Patients who have never received virtual reality therapy
7. Upper extremity Brunnstrom Stage III and above
8. Patients with a spasticity level below 3 according to the Modified Ashworth Scale (MAS) in the affected upper extremity (MAS 1-5 rating system)
9. Patients who agreed to participate in the study and signed the informed consent form

Exclusion Criteria:

1. History of seizures or epilepsy (except childhood febrile seizures),
2. Arthritis or pain in the affected upper limb that limits repetitive exercise,
3. Severe aphasia, cognitive impairment (premorbid dementia) or psychiatric disorders,
4. Spasticity in the affected arm is 3 or more compared to MAS,
5. Patients without sitting balance,
6. Patients with posterior cerebral artery infarction,
7. Patients with subarachnoid hemorrhage,
8. Patients with visual impairments that may affect the virtual reality application

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Post-stroke patients consecutively admitted to Ankara University Faculty of Medicine, Department of Physical Medicine and Rehabilitation will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-06-22 (Actual); Primary Completion 2026-06-22 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
The feasibility of using BeCureTM virtual reality in stroke patients will be determined according to the System Usability Scale (SUS) score. | Baseline and 7 days
  The System Usability Scale (SUS) is a simple, ten-item Likert scale of subjective evaluations of usability. It was developed in 1986 by John Brooke for usability evaluation. In short, it is a standardized questionnaire to measure users' satisfaction with a product or system. At the same time, a score between 0-100 can be obtained with SUS. When calculating the exact score, 1 is subtracted from the given value of items 1, 3, 5, 7 and 9 (odd numbered and positive opinion). The scores for items 2, 4, 6, 8 and 10 (items with negative opinions) are subtracted from 5. The SUS score can then be found by adding them all together and multiplying this sum by 2.5 to complete the 0-100 range. The minimum score is 0 points and the maximum score is 100 points. A higher score indicates better usability.

SECONDARY OUTCOMES:
1- A patient feedback questionnaire on the safety of BeCureTM virtual reality use will be completed. | Baseline and 7 days
  1. Patient feedback questionnaire will be completed for the reliability of BeCureTM virtual reality use in stroke patients.
  2. The relationship between the use of BeCureTM virtual reality and cognitive functions in stroke patients will be determined by the Montreal Cognitive Assessment Scale and Mini Mental State Examination.

CONTACTS AND LOCATIONS:
Overall Officials: Sehim Kutlay, Professor, Study Director — Ankara University
Locations (1):
- Ankara University School of Medicine Department of Physical Medicine and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided